CLINICAL TRIAL: NCT04636502
Title: Subcutaneous Immune Globulin (SCIG 20%) and Facilitated Subcutaneous Immunoglobulin (fSCIG) Treatment in Polish Paediatric Patients With Primary Immunodeficiencies (PID) - Retrospective Medical Chart Review Study
Brief Title: Retrospective, Observational Chart Review Study Conducted in Poland to Document the Management and Clinical Outcome of CUVITRU and HYQVIA in Pediatric Participants (< 18 Years) With Primary Immunodeficiency (PID)
Acronym: IG-TATRY
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: PID-4001
Record Dates: First submitted 2020-11-18; First posted 2020-11-19 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Primary Immunodeficiencies (PID)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort: Participants who had treated with fSCIG (HyQvia) for not more than 27 months and SCIG 20% (Cuvitru) for not more than 35 months.

SUMMARY:
The purpose of this observational, multi-center, retrospective cohort study is to assess treatment patterns of Cuvitru (SCIG) 20 percent (%) and HyQvia (fSCIG) in polish pediatric participants with PID. The study will collect pediatric patient data. These data are gathered and collected during routine clinical care. As this is a non-interventional/observational study, no treatment/pharmacotherapy is provided as part of the study.

DETAILED DESCRIPTION:
Subcutaneous immune globulin (SCIG 20%) and facilitated subcutaneous immunoglobulin (fSCIG) treatment in Polish paediatric patients with primary immunodeficiencies (PID) - retrospective medical chart review study

ELIGIBILITY:
Inclusion Criteria:

Participant eligibility is determined according to the following criteria prior to entry into the study:

* The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
* Male or female participants with PID, aged less than (<)18 years treated with SCIG 20% or fSCIG..
* Diagnosis of PID according to the criteria developed by the European Society for Immunodeficiencies (ESID) https://esid.org/About-ESID
* Treatment period for 20% SCIG ranges from November 1, 2017 until June 30, 2020, and for fSCIG from July 1, 2018 until June 30, 2020.

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants with PID on treatment with SCIG 20% or fSCIG will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Number of Doses per Infusion | From start of the study upto end of the study (6 months)
Number of Infusion Sites | From start of the study upto end of the study (6 months)
Infusion Volume | From start of the study upto end of the study (6 months)
Method of Administration | From start of the study upto end of the study (6 months)
  Method of administration in participants will be through pump or rapid push.
Length of Needle | From start of the study upto end of the study (6 months)
  Length of needle used for infusions will be assessed.
Assessment of Person who Perform the Infusion | From start of the study upto end of the study (6 months)
  Assessment of person (parent/guardian or self) who performs the infusion will be assessed.
Type of Pump | From start of the study upto end of the study (6 months)
Total Dose per 4 weeks | From start of the study upto end of the study (6 months)
  Total dose administered per 4 weeks data will be assessed.
Total Infusion Volume per 4 Weeks | From start of the study upto end of the study (6 months)
Treatment Interval per 4 Weeks | From start of the study upto end of the study (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (5):
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytecki Szpital Dziecięcy w Krakowie, Krakow
  - Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw
  - Wojewódzki Szpital Specjalistyczny im. J. Gromkowskiego, Wroclaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. prof. Stanisława Szyszko Śląskiego Uniwersytetu Medycznego w Katowicach, Zabrze

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Mach-Tomalska M, Pituch-Noworolska A, Bien E, Malanowska M, Machura E, Pukas-Bochenek A, Chrobak E, Pac M, Pietrucha B, Drygala S, Kamieniak M, Kasprzak J, Heropolitanska-Pliszka E. Facilitated subcutaneous immunoglobulin treatment patterns in pediatric patients with primary immunodeficiency diseases. Immunotherapy. 2024 Apr;16(6):391-403. doi: 10.2217/imt-2023-0305. Epub 2024 Feb 16. PMID 38362629
- [Derived] Heropolitanska-Pliszka E, Pac M, Pietrucha B, Machura E, Pukas-Bochenek A, Chrobak E, Bien E, Malanowska M, Pituch-Noworolska A, Drygala S, Kamieniak M, Kasprzak J, Mach-Tomalska M. Subcutaneous immunoglobulin 20% (Ig20Gly) treatment regimens in pediatric patients with primary immunodeficiencies - real-world data from the IG TATRY study. Expert Rev Clin Immunol. 2023 Jul-Dec;19(10):1281-1291. doi: 10.1080/1744666X.2023.2240514. Epub 2023 Jul 25. PMID 37489744
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5fb63601d98d000029649dce